CLINICAL TRIAL: NCT02273141
Title: A Multicenter Randomized Parallel Group Phase III Study Comparing the Bowel Cleansing Efficacy, Safety and Tolerability of NER1006 (a Low Volume Bowel Cleansing Solution) Versus Sodium Picosulfate and Magnesium Salt (SP+MS) Solution Using Day Before-Only Dosing Regimen in Adults.
Brief Title: Multicenter Randomized Parallel Group Phase III Study Comparing the Bowel Cleansing Efficacy, Safety and Tolerability of NER1006 Versus a Sodium Picosulfate and Magnesium Salt Solution Using Day Before-Only Dosing Regimen in Adults.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: NER1006-03/2014 (DAYB)
Record Dates: First submitted 2014-10-16; First posted 2014-10-23 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-04

CONDITIONS: Colorectal Cancer; Colorectal Carcinoma; Colon Cleansing
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NER1006, Day Before-Only Dosing (Experimental): NER1006 1-Day Day Before-Only Split-Dosing Regimen (to commence on the evening of the day before colonoscopy).
  Interventions: Drug: NER1006, Day Before-Only Dosing
- SP+MS, Day Before-Only Dosing (Active Comparator): SP+MS 1-Day Day Before-Only Split-Dosing Regimen (to commence on the morning of the day before colonoscopy).
  Interventions: Drug: SP+MS, Day Before-Only Dosing

INTERVENTIONS:
Drug: NER1006, Day Before-Only Dosing — The subject will self-administer both doses of NER1006 in the evening of Day 1 with 1-2 hours interval. Subject will take mandatory additional clear fluid after each dose.
  Arms: NER1006, Day Before-Only Dosing
Drug: SP+MS, Day Before-Only Dosing — The subject will self-administer SP+MS in the morning of Day 1 and afternoon of Day 1. Subject will take mandatory additional clear fluid after each dose.
  Arms: SP+MS, Day Before-Only Dosing

SUMMARY:
This study evaluates the efficacy, safety and tolerability of NER1006 versus a sodium picosulfate and magnesium salt solution (SP + MS) in adult patients requiring bowel cleansing prior to any procedure that requires a clean bowel, using a Day Before Only Dosing regimen. Approximately 484 patients will be randomised with the aim of achieving a minimum of 220 patients in each of the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent.
* Male and female outpatients and inpatients aged: ≥18 to ≤85 years undergoing a screening, surveillance or diagnostic colonoscopy.
* Females of child-bearing potential must have a negative pregnancy test at Screening and at Visit 2 and must be practising one of the following methods of birth control and agree to continue with the regimen throughout the study period (unless postmenopausal or surgically sterile, or whose sole sexual partner has had a successful vasectomy):

  * Oral, implantable, or injectable contraceptives (for a minimum of three months before study entry) in combination with a condom;
  * Intrauterine device in combination with a condom;
  * Double barrier method (condom* and occlusive cap [diaphragm or cervical/vault caps] with spermicidal foam/gel/film/cream/suppository).
* Willing, able and competent to complete the entire study and to comply with instructions.

Exclusion Criteria:

* Patients with past history within last 12 months or current episode of severe constipation (requiring repeated use of laxatives/enema or physical intervention before resolution), known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or megacolon.
* Patients with ongoing severe acute Inflammatory Bowel Disease.
* Patients who have had previous significant gastrointestinal surgeries, including colonic resection, sub-total colectomy, abdomino-perineal resection, de-functioning colostomy, Hartmann's procedure and de-functioning ileostomy or other similar surgeries involving structure and function of the small or large colon.
* Regular use of laxatives or colon motility altering drugs in the last month (i.e. more than 2-3 times per week) and/or laxative use within 72 hours prior to administration of the preparation.
* Patients with active intestinal bleeding episodes or with a clinically significant low hemoglobin level <9 g/dL for women and <11 g/dL for men at screening.
* Known glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Known phenylketonuria.
* Known hypersensitivity to polyethylene glycols, ascorbic acid and sulfates (not including sulfa-based products), sodium picosulfate and magnesium salt compounds, or any other component of the study drug or comparator
* Past history within the last 12 months or evidence of any on-going clinically relevant electrocardiogram abnormalities (e.g. arrhythmias).
* History of uncontrolled hypertension with systolic blood pressure >170 mmHg and diastolic blood pressure >100 mmHg.
* Patients with cardiac insufficiency NYHA grades III or IV.
* Patients with moderate to severe renal insufficiency (i.e. with GFR, <60 mL/min/1.73m2).
* Patient with serum albumin <3.4 g/dL.
* Patients with liver disease of grades B and C according to the Child Pugh classification.
* Patients suffering from dehydration at screening as evaluated by the Investigator from physical examination and laboratory investigations.
* Patients with clinically significant electrolyte abnormalities, whether pre-existing or noted at screening, such as hypernatremia, hyponatremia, hyperphosphatemia, hypermagnesemia, hypokalemia, hypocalcaemia, dehydration, or those secondary to the use of diuretics or angiotensin converting enzyme (ACE) inhibitors.
* Patients with any other clinically significant hematological parameters including coagulation profile at screening.
* Patients with impaired consciousness that might predispose them to pulmonary aspiration.
* Patients undergoing colonoscopy for foreign body removal and/or decompression.
* Patients who are pregnant or lactating, or intending to become pregnant during the study.
* Clinically relevant findings on physical examination based on the Investigator's judgment.
* History of drug or alcohol abuse within the 12 months prior to dosing.
* Concurrent participation in an investigational drug or device study or participation within three months of study entry.
* Patients who are ordered to live in an institution on court or authority order.
* Patients with history of rhabdomyolysis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schreiber, Principal Investigator — University Hospital Schleswig-Holstein
Locations (19):
- Germany (3):
  - Charité - Campus Virchow Klinikum, Berlin
  - University Hospital Schleswig-Holstein, Kiel
  - An der Germania Brauerei 6, Münster
- Italy (3):
  - An der Germania Brauerei 6, Milan
  - Osp.San Raffaele U.O. Gastroenterologia, Milan
  - P.T.P.Nuovo Regina Margherita, Rome
- Netherlands (4):
  - Onze Lieve Vrouwe Gashuis, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Radboud UMC, Nijmegen
  - Orbis Medisch Centrum, Sittard
- Poland (4):
  - Centrum Medyczne sw. Lukasza, Częstochowa
  - Instytut Medycyny Wsi im. Witolda Chodzki w, Lubliniec
  - Specjalistyczna Praktyka Lekarska dr med. Marek Horynski, Sopot
  - SPSK Nr 1 im. Prof. Tadeusza Sokolowskiego, Szczecin
- Spain (3):
  - Hospital de Vinalopó, Unidad de Endoscopia Digestiva, Elche
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario La Paz, Unidad Enfermedad Intestinal, Madrid
- United Kingdom (2):
  - Department of Surgery, Raigmore Hospital, Inverness
  - Derriford Hospital, Plymouth

REFERENCES:
- [Derived] Cash BD, Allen C, Poppers DM. Transient alterations in plasma sodium concentrations with NER1006 bowel preparation: an analysis of three phase III, randomized clinical trials. BMC Gastroenterol. 2022 Sep 5;22(1):412. doi: 10.1186/s12876-022-02484-7. PMID 36064325

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial recruited out/in-patients at 19 medical centres in Europe, from November 2014 to July 2015.
Period: Overall Study
Arm/Group | SP+MS, Day Before-Only Dosing | NER1006, Day Before-Only Dosing
Started | 257 | 258
Completed | 240 | 233
Not Completed | 17 | 25
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 10 | 15
Not completed — Various | 6 | 6

BASELINE CHARACTERISTICS:
Population: The number of participants for analysis, 220 per arm, was based on assumed overall cleansing success rates of 70% for SP+MS and 75% for NER1006, a non-inferiority margin of 10%, and at least 90% power to demonstrate non-inferiority. The overall number of participants analyzed was based on the modified full analysis set (mFAS).
Groups:
- SP+MS, Day Before-Only Dosing: SP+MS 1-Day Day Before-Only Split-Dosing Regimen (to commence on the moring of the day before colonoscopy).
- Total: Total of all reporting groups
Arm/Group | SP+MS, Day Before-Only Dosing | NER1006, Day Before-Only Dosing | Total
Number analyzed (Participants) | 257 | 258 | 515
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 207 | 203 | 410
  >=65 years | 50 | 54 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (13.35) | 54.6 (11.64) | 53.8 (12.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 168 | 342
  Male | 83 | 90 | 173

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Successful Bowel Cleansing (Overall Colon)
Description: The overall quality of bowel cleansing was assessed by a blinded central reader (an experienced and trained colonoscopist) using the segmental scores of the Harefield Cleansing Scale (HCS). A final HCS grading of A, B, C or D was derived. Grades A and B are classified as successful (i.e. all mucosa could be visualized) and C and D are classified as unsuccessful. Comparison of overall success of cleansing with NER1006 versus SP+MS was evaluated using a non-inferiority study design.
Time Frame: One day (day before colonoscopy)
Population: The overall number of participants analyzed was based on the mFAS. This included all randomized patients, except any patient who (i) was randomized but subsequently failed to meet entry criteria and (ii) in whom it was confirmed (from their patient diary) that the same patient did not receive any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | SP+MS, Day Before-Only Dosing | NER1006, Day Before-Only Dosing
Number analyzed (Participants) | 251 | 250
Participants
  Successful | 135 | 155
  Failure | 116 | 95
Statistical Analysis 1: Comparison: SP+MS, Day Before-Only Dosing vs NER1006, Day Before-Only Dosing; The hypothesis was to demonstrate non-inferiority (NI) of NER1006 regimen to SP+MS (10% margin). Success rate was no. of patients with successful overall bowel cleansing as proportion of no. of patients in each group. Treatment effect was NER1006 success rate - SP+MS success rate. A Hochberg procedure was used to control Type I error since there were 2 alternative primary endpoints. An alpha level of 1.25% 1-sided was used. A closed testing procedure used to evaluate superiority if NI was met; Test type: Non-Inferiority or Equivalence — The confidence limits were adjusted for multiple comparisons (two alternative primary endpoints): To be declared non-inferior, the primary endpoint must show a difference in success rates of no greater than 10% in favor of SP+MS using lower 1-sided 97.5% confidence limits. Calculated using exact Clopper-Pearson confidence limits; p = 0.038, Fisher Exact — The p-value was adjusted for multiple comparisons (2 alternative primary endpoints): To be declared superior, the primary endpoint must demonstrate non-inferiority with 1-sided p-value <0.025, the threshold for statistical significance; Difference in success rate = 8.22, 97.5% CI 1-sided [lower limit -0.50]

2. Primary Outcome: Number of Patients With 'Excellent Plus Good' (Highly Effective) Bowel Cleansing (Colon Ascendens)
Description: The overall quality of bowel cleansing was assessed by a blinded central reader (an experienced and trained colonoscopist) using the segmental scores of the Harefield Cleansing Scale (HCS). Highly effective cleansing in the colon ascendens corresponded to scores 3 (Good) or 4 (Excellent) of the HCS. Adequate plus failure of cleansing corresponded to score 0-2. Comparison of 'Excellent plus good' cleansing of the colon ascendens using NER1006 versus SP+MS was evaluated using a non-inferiority study design.
Time Frame: One day (day before colonoscopy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SP+MS, Day Before-Only Dosing | NER1006, Day Before-Only Dosing
Number analyzed (Participants) | 251 | 250
Participants
  Excellent plus good | 3 | 11
  Adequate plus failure | 248 | 239
Statistical Analysis 1: Comparison: SP+MS, Day Before-Only Dosing vs NER1006, Day Before-Only Dosing; Hypothesis was to demonstrate NI of NER1006 regimen to SP+MS (10% margin). Success rate was no. of patients with highly effective cleansing of the colon ascendens as proportion of no. of patients in each group. Treatment effect was NER1006 success rate - SP+MS success rate. A Hochberg procedure was used to control Type I error since there were 2 alternative primary endpoints. An alpha level of 1.25% 1-sided was used. A closed testing procedure used to evaluate superiority if NI was met; Test type: Non-Inferiority or Equivalence — The confidence limits were adjusted for multiple comparisons (two alternative primary endpoints): To be declared non-inferior the primary endpoint must show a difference in success rates of no greater than 10% in favor of SP+MS using lower 1-sided 97.5% confidence limits. Calculated using exact Clopper-Pearson confidence limits; p = 0.027, Fisher Exact — The p-value was adjusted for multiple comparisons (2 alternative primary endpoints): To be declared superior, primary endpoint must demonstrate non-inferiority with 1-sided p-value <0.025, the threshold for statistical significance; Difference in excellent plus good rate = 3.20, 97.5% CI 1-sided [lower limit -5.56]

3. Secondary Outcome: Adenoma Detection Rate (Colon Ascendens)
Description: Comparison of the number of patients with at least one adenoma detected in the colon ascendens when NER1006 is used for bowel cleansing versus SP+MS. Adenoma detection rate (ADR) defined as the number of patients with at least one adenoma in the colon ascendens.
Time Frame: One day (day before colonoscopy).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SP+MS, Day Before-Only Dosing | NER1006, Day Before-Only Dosing
Number analyzed (Participants) | 251 | 250
Participants
  Patients with no adenomas detected | 241 | 234
  Patients with at least one adenoma detected | 10 | 16
Statistical Analysis 1: Comparison: SP+MS, Day Before-Only Dosing vs NER1006, Day Before-Only Dosing; If at least one of the alternative primary endpoints was met, then key secondary endpoints for the same colon region as met by the primary endpoint were evaluated hierarchically in a pre-specified order. The difference in ADR was calculated as NER1006 rate - SP+MS rate using 1-sided 97.5% confidence limits. Formal testing was to proceed in the hierarchy if preceding key secondary endpoint met non-inferiority. This procedure ensured overall Type I error control at 2.5% 1-sided; Test type: Non-Inferiority or Equivalence — To be declared non-inferior, the key secondary endpoint must show a difference in rates of no greater than 10% in favor of SP+MS using lower 1-sided 97.5% confidence limits. Calculated using exact Clopper-Pearson confidence limits; p = 0.154, Fisher Exact — To be declared superior, the key secondary endpoint must demonstrate non-inferiority and show a significant advantage for NER1006 relative to SP+MS with 1-sided p-value <0.025, the threshold for statistical significance; Difference in ADR = 2.42, 95% CI 2-sided [-6.35 to 11.12]

4. Secondary Outcome: Adenoma Detection Rate (Overall Colon)
Description: Comparison of the number of patients with at least one adenoma detected in the overall colon when NER1006 is used for bowel cleansing versus SP+MS. Adenoma detection rate (ADR) defined as the number of patients with at least one adenoma in the overall colon.
Time Frame: One day (day before colonoscopy)
Population: The overall number of participants analyzed was based on the mFAS. This included all randomized patients with the exception of any patient who was randomized but subsequently failed to meet entry criteria and in whom it was confirmed (from their patient diary) that the same patient did not receive any study drug (n=501).
Measure: Count of Participants; unit: Participants
Arm/Group | SP+MS, Day Before-Only Dosing | NER1006, Day Before-Only Dosing
Number analyzed (Participants) | 251 | 250
Participants
  Patients with no adenomas detected | 204 | 195
  Patients with at least one adenoma detected | 47 | 55
Statistical Analysis 1: Comparison: SP+MS, Day Before-Only Dosing vs NER1006, Day Before-Only Dosing; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.212, Fisher Exact — [p-value comment as in outcome 3, analysis 1]; Difference in ADR = 3.27, 95% CI 2-sided [-5.56 to 11.91]

5. Secondary Outcome: Polyp Detection Rate (Colon Ascendens)
Description: Comparison of the number of patients with at least one polyp detected in the colon ascendens when NER1006 is used for bowel cleansing versus SP+MS. Polyp detection rate (PDR) defined as the number of patients with at least one polyp in the colon ascendens.
Time Frame: One day (day before colonoscopy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SP+MS, Day Before-Only Dosing | NER1006, Day Before-Only Dosing
Number analyzed (Participants) | 251 | 250
Participants
  Patients with no polyps detected | 232 | 220
  Patients with at least one polyp detected | 19 | 30
Statistical Analysis 1: Comparison: SP+MS, Day Before-Only Dosing vs NER1006, Day Before-Only Dosing; If at least one of the alternative primary endpoints was met, then key secondary endpoints for the same colon region as met by the primary endpoint were evaluated hierarchically in a pre-specified order. The difference in PDR was calculated as NER1006 rate - SP+MS rate using 1-sided 97.5% confidence limits. Formal testing was to proceed in the hierarchy if preceding key secondary endpoint met non-inferiority. This procedure ensured overall Type I error control at 2.5% 1-sided; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.064, Fisher Exact — [p-value comment as in outcome 3, analysis 1]; Difference in PDR = 4.43, 95% CI 2-sided [-4.36 to 13.10]

6. Secondary Outcome: Polyp Detection Rate (Overall Colon)
Description: Comparison of the number of patients with at least one polyp detected in the overall colon when NER1006 is used for bowel cleansing versus SP+MS. Polyp detection rate (PDR) defined as the number of patients with at least one polyp in the overall colon.
Time Frame: One day (day before colonoscopy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SP+MS, Day Before-Only Dosing | NER1006, Day Before-Only Dosing
Number analyzed (Participants) | 251 | 250
Participants
  Patients with no polyps detected | 160 | 152
  Patients with at least one polyp detected | 91 | 98
Statistical Analysis 1: Comparison: SP+MS, Day Before-Only Dosing vs NER1006, Day Before-Only Dosing; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.278, Fisher Exact — [p-value comment as in outcome 3, analysis 1]; Difference in PDR = 2.95, 95% CI 2-sided [-5.96 to 11.51]

ADVERSE EVENTS:
Time Frame: Morning of Day 1 (first dose) to Day 9 (final clinic visit)
Description: Safety analyses were based on the safety population which included all randomized patients for whom it could not be ruled out (from their patient diary) that they received study drug at least once (n=476). The analyses are based on treatment emergent adverse events (TEAEs). There were no deaths and the serious TEAE was not related to treatment.
Arm/Group | SP+MS, Day Before-Only Dosing | NER1006, Day Before-Only Dosing
All-Cause Mortality (participants affected / at risk) | 0/241 | 0/235
Serious Adverse Events (participants affected / at risk) | 0/241 | 1/235
Other Adverse Events (participants affected / at risk) | 9/241 | 32/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SP+MS, Day Before-Only Dosing (N=241) | NER1006, Day Before-Only Dosing (N=235)
Ovarian abscess (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SP+MS, Day Before-Only Dosing (N=241) | NER1006, Day Before-Only Dosing (N=235)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 8 (8)
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 11 (11)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 4 (5)

LIMITATIONS AND CAVEATS:
Imputation of failure occurred in 4% of patients. This strict analytical approach reduced the cleansing success rates for both treatments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No